CLINICAL TRIAL: NCT06777771
Title: The Effects of Reformer Pilates on Pain, Functional Capacity, Lumbopelvic Stabilization, Abdominal Muscles, Respiratory Functions, Pelvic Floor Function, and Venous Insufficiency in Pregnant Women
Brief Title: Effects of Reformer Pilates in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Assoc. Prof., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Reformer pilates in pregnancy
Record Dates: First submitted 2024-12-27; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Pelvic Floor Disorders; Pain, Back; Pain, Neck; Pregnancy, Abdominal
Keywords: Pregnancy; Exercise; Reformer Pilates; Pilates; Pelvic Floor Dysfunction; Lumbopelvic Stabilization; Functional Capacity; Respiratory Function; Abdominal Muscle Thickness; Venous Insufficiency; Urinary Incontinence; Sexual Function; Pain
MeSH Terms: conditions — Pelvic Floor Disorders; Back Pain; Neck Pain; Pregnancy, Abdominal; Motor Activity; Respiratory Aspiration; Venous Insufficiency; Urinary Incontinence; Pain

STUDY DESIGN:
Intervention Model Description: Exercise group and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Reformer pilates sessions will be applied to the participants in the exercise group.
  Interventions: Other: Reformer pilates exercises
- Control group (No Intervention): Participants in the control group will be recommended to walk.

INTERVENTIONS:
Other: Reformer pilates exercises — The reformer pilates exercises session will start with 5 minutes of warm-up exercises, continue with resistance exercises for 20 minutes, and end with 5 minutes of cool-down exercises. The springs of the reformer pilates device will be adjusted to create mild fatigue in the first week and will be gradually increased to create moderate fatigue in the following weeks. Reformer pilates sessions will consist of 15-20 different exercises with 12-15 repetitions, including all major muscle groups. These sessions will also include exercises that strengthen the pelvic floor muscles. Reformer pilates sessions will be applied twice a week for 6 weeks, a total of 12 sessions. Apart from this, they will be asked to walk for at least 30 minutes a day, at least 3 days a week.
  Arms: Exercise group

SUMMARY:
Pregnancy is known as a period associated with important physiological and psychological changes in women's lives. There is moderately sufficient evidence in the literature to recommend supplementing prenatal physical activity for maternal health benefits. It has been reported that physical exercise by pregnant women in the absence of obstetric contraindications will not pose a risk to the health of the mother and fetus. In the literature, there are no studies examining the effects of reformer pilates on pain, functional capacity, lumbopelvic stabilization, diastasis recti abdominis, abdominal muscle thickness, respiratory functions, pelvic floor dysfunction, urinary incontinence, sexual function, and venous insufficiency in pregnant women. Therefore, this study aimed to investigate the effects of reformer pilates on pain, functional capacity, lumbopelvic stabilization, diastasis recti abdominis, abdominal muscle thickness, respiratory functions, pelvic floor dysfunction, urinary incontinence, sexual function, and venous insufficiency in pregnant women.

DETAILED DESCRIPTION:
Pregnancy is one of the most serious periods in a woman's life and lasts approximately forty weeks. Many anatomical, physiological, and psychological changes occur in pregnant women. The main reasons for these are hormonal changes, increase in total blood volume, growth of the uterus, and postural changes due to the shift of the body's center of gravity.

Even though the etiology and pathogenesis of low back pain occurring during pregnancy have not been clearly explained, it is assumed to be multifactorial. Low back pain during pregnancy is common and affects approximately half of pregnant women. Additionally, pain may occur in the low back and sacroiliac joints due to postural changes that occur with the growth of the fetus. Low back pain and pelvic girdle pain are among the most common musculoskeletal complaints in pregnant women.

Studies conducted on pregnant women and women in the postpartum period have reported changes in the length, thickness, and separation amount of the abdominal muscles and the morphological features of the rectus abdominis muscle.

The strength and thickness of the pelvic floor muscles may decrease in pregnant women. Pregnancy and birth are major risk factors for urinary incontinence. Additionally, a relationship between pregnancy and sexual dysfunction has been reported in the literature.

To meet the needs of the fetus during pregnancy, changes occur in many organs and systems, as well as changes in the uterus. One of these is the adaptation seen in the respiratory system. Another change is the adaptation in the venous system. Pregnancy is one of the factors that increase the risk of developing venous insufficiency.

Pregnancy is known as a period associated with important physiological and psychological changes in women's lives. Pregnancy and exercise are biological processes. These cause many adaptations in the body, which may be in the same or the opposite direction. There is moderately sufficient evidence in the literature to recommend promoting prenatal physical activity for maternal health benefits.

In the literature, no study has been found investigating the effects of reformer pilates on pain, functional capacity, lumbopelvic stabilization, diastasis recti abdominis, abdominal muscle thickness, respiratory functions, pelvic floor dysfunction, urinary incontinence, sexual function, and venous insufficiency in pregnant women. For this reason, this study aimed to investigate the effects of reformer pilates on pain, functional capacity, lumbopelvic stabilization, diastasis recti abdominis, abdominal muscle thickness, respiratory functions, pelvic floor dysfunction, urinary incontinence, sexual function, and venous insufficiency in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Primiparous pregnancy
* Adult pregnant women (between 18-35 years old)
* Pregnant women whose gestational week is 11-22 weeks
* Pregnant women with a body mass index <30
* Ability to read and write

Exclusion Criteria:

* Multiple pregnancies
* Having a history of abdominal surgery
* Having one of the conditions in which exercise is contraindicated, such as heart disease, severe lung disease, continuous bleeding in the second and third trimesters, placenta previa, risk of premature birth, rupture of membranes, preeclampsia, severe anemia
* Not volunteering to participate in the study
* Not participating in more than 90% of the training sessions

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Thickness measurement of the rectus abdominis muscle | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The thickness of the rectus abdominis muscle will be measured approximately 4 cm lateral to the umbilicus using a 2-7 MHz linear probe (Voluson E8, General Electrics, USA) while participants are lying in a supine position. The measurement will be repeated 3 times, and the average will be recorded in millimeters. The measurements to be made with USG will be made unilaterally by a specialist physician during axial imaging.
Thickness measurement of the transversus abdominis muscle | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The thickness of the transversus abdominis muscle will be measured at the intersection point of the umbilicus and axillary line using a 2-7 MHz linear probe (Voluson E8, General Electrics, USA) while participants are lying in a supine position. The measurement will be repeated 3 times, and the average will be recorded in millimeters. The measurement to be made with USG will be made unilaterally by a specialist physician during axial imaging.
Thickness measurement of the external oblique abdominal muscle | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The thickness of the external oblique abdominal muscle will be measured at the intersection point of the umbilicus and axillary line using a 2-7 MHz linear probe (Voluson E8, General Electrics, USA) while participants are lying in a supine position. The measurement will be repeated 3 times, and the average will be recorded in millimeters. The measurement to be made with USG will be made unilaterally by a specialist physician during axial imaging.
Thickness measurement of the internal oblique abdominal muscle | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The thickness of the internal oblique abdominal muscle will be measured at the intersection point of the umbilicus and axillary line using a 2-7 MHz linear probe (Voluson E8, General Electrics, USA) while participants are lying in a supine position. The measurement will be repeated 3 times, and the average will be recorded in millimeters. The measurement to be made with USG will be made unilaterally by a specialist physician during axial imaging.
The forced vital capacity (FVC) value | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The forced vital capacity (FVC) value will be measured with a spirometric test using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. During the test, participants will be asked to take a deep breath and then release it as much as possible until there is no air left in their lungs. The test will be repeated 3 times. The average of the two best test results will be recorded.
The forced expiratory volume in the first second (FEV1) value | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The forced expiratory volume in the first second (FEV1) value will be measured with a spirometric test using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. During the test, participants will be asked to take a deep breath and then release it as much as possible until there is no air left in their lungs. The test will be repeated 3 times. The average of the two best test results will be recorded.
The forced expiratory volume in the first second (FEV1)/the forced vital capacity (FVC) (FEV1/FVC) value | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The forced expiratory volume in the first second (FEV1)/the forced vital capacity (FVC) (FEV1/FVC) value will be measured with a spirometric test using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. During the test, participants will be asked to take a deep breath and then release it as much as possible until there is no air left in their lungs. The test will be repeated 3 times. The average of the two best test results will be recorded.
The peak expiratory flow (PEF) value | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The peak expiratory flow (PEF) value will be measured with a spirometric test using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. During the test, participants will be asked to take a deep breath and then release it as much as possible until there is no air left in their lungs. The test will be repeated 3 times. The average of the two best test results will be recorded.
Pelvic Floor Dysfunction Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants' pelvic floor dysfunction value will be assessed using the Pelvic Floor Distress Inventory-20 (PTDE-20). The total score that may be obtained from the PTDE-20 ranges from "0" (best score) to "300" (worst score). High scores indicate higher levels of pelvic floor dysfunction.

SECONDARY OUTCOMES:
Neck Pain Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The presence of neck pain will be recorded as "present" or "absent". In the case of pain, the pain intensity will be measured using the Visual Analogue Scale (VAS). In addition, the duration and frequency of pain and activities that reduce or increase pain will be questioned.
Back Pain Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The presence of back pain will be recorded as "present" or "absent". In the case of pain, the pain intensity will be measured using the Visual Analogue Scale (VAS). In addition, the duration and frequency of pain and activities that reduce or increase pain will be questioned.
Low Back Pain Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The presence of low back pain will be recorded as "present" or "absent". In the case of pain, the pain intensity will be measured using the Visual Analogue Scale (VAS). In addition, the duration and frequency of pain and activities that reduce or increase pain will be questioned.
Pelvic Girdle Pain Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The presence of pelvic girdle pain will be recorded as "present" or "absent". In the case of pain, the intensity of pain in that area will be measured using the Visual Analogue Scale (VAS). In addition, the duration and frequency of pain and activities that reduce or increase pain will be questioned.
Functional Capacity Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  The functional capacity level of the participants will be evaluated with the five-repetition sit-to-stand test. Participants will be asked to get up and sit down 5 times as quickly as possible. This test will be applied 2 times and the average value will be taken.
Lumbopelvic Stabilization Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants' lumbopelvic stabilization level will be evaluated in the supine position using a pressure-stabilizing feedback device (Pressure Biofeedback Unit, Chattanooga Group, Hixon, TN, USA). The pressure will be adjusted to 40 mmHg. During the test, the abdominal muscles will contract isometrically to keep the lumbar region and pelvis stable, while the load is gradually added with lower extremity movements so that the pressure remains constant. In this test, which consists of five levels, the load acting on the lumbopelvic region is increased with lower extremity movements while progressing from the first level to the fifth level.
Urinary Incontinence Severity Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants' urinary incontinence severity level will be assessed using the Incontinence Severity Index (ISI). A score between 1 and 12 is taken from the ISI. High scores indicate higher urinary incontinence severity.
Sexual Function Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants' sexual function level will be assessed using the Female Sexual Function Index (FSFI). The highest score that may be obtained from the FSFI is 36 and the lowest score is 2. If the score is above 26.5, it means that the sexual function is normal. Values below 26.5 indicate sexual dysfunction.
Diastasis Recti Abdominis Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants will be placed in the supine position. The practitioner's fingers will be vertically on the linea alba. The participant will be asked to raise their head and shoulders off the ground while extending their arms forward. During the measurement, the amount of separation of the two parts of the rectus abdominis muscle will be recorded as the centimeter value of the fingers between the two parts of this muscle. This measurement will be made from the umbilicus, 8-10 cm below and above the umbilicus along the linea alba.
Venous Insufficiency Assessment | First evaluation (baseline) and final evaluation (6 weeks after first evaluation)
  Participants' venous insufficiency status will be evaluated with the clinical classification subheading of the CEAP classification.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Prof.Dr., Study Director — Izmir Democracy University; Kübra Özonay, PhD student, Principal Investigator — Izmir Democracy University
Locations (1):
- İzmir Democracy Univercity, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilchinsky T, Tene L, Kalichman L. Pilates exercises during pregnancy: A narrative review. J Bodyw Mov Ther. 2024 Oct;40:1146-1152. doi: 10.1016/j.jbmt.2024.07.038. Epub 2024 Jul 18. PMID 39593426
- [Background] Ferraz VS, Peixoto C, Ferreira Resstel AP, Cerqueira de Paula YT, Gomes de Souza Pegorare AB. Effect of the pilates method on pain and quality of life in pregnancy: A systematic review and meta-analysis. J Bodyw Mov Ther. 2023 Jul;35:220-227. doi: 10.1016/j.jbmt.2023.04.076. Epub 2023 May 3. PMID 37330773
- [Background] Mazzarino M, Kerr D, Morris ME. Feasibility of pilates for pregnant women: A randomised trial. J Bodyw Mov Ther. 2022 Oct;32:207-212. doi: 10.1016/j.jbmt.2022.05.001. Epub 2022 May 8. PMID 36180151
- [Background] Von Aarburg N, Veit-Rubin N, Boulvain M, Bertuit J, Simonson C, Desseauve D. Physical activity and urinary incontinence during pregnancy and postpartum: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2021 Dec;267:262-268. doi: 10.1016/j.ejogrb.2021.11.005. Epub 2021 Nov 16. PMID 34839247
- [Background] Chan CWH, Au Yeung E, Law BMH. Effectiveness of Physical Activity Interventions on Pregnancy-Related Outcomes among Pregnant Women: A Systematic Review. Int J Environ Res Public Health. 2019 May 23;16(10):1840. doi: 10.3390/ijerph16101840. PMID 31126153
- [Background] Rodriguez-Diaz L, Ruiz-Frutos C, Vazquez-Lara JM, Ramirez-Rodrigo J, Villaverde-Gutierrez C, Torres-Luque G. Effectiveness of a physical activity programme based on the Pilates method in pregnancy and labour. Enferm Clin. 2017 Sep-Oct;27(5):271-277. doi: 10.1016/j.enfcli.2017.05.008. Epub 2017 Jul 6. English, Spanish. PMID 28689647
- [Background] Benjamin DR, van de Water AT, Peiris CL. Effects of exercise on diastasis of the rectus abdominis muscle in the antenatal and postnatal periods: a systematic review. Physiotherapy. 2014 Mar;100(1):1-8. doi: 10.1016/j.physio.2013.08.005. Epub 2013 Oct 5. PMID 24268942